CLINICAL TRIAL: NCT00666588
Title: A Phase II Pilot Study of Bortezomib (PS-341, Velcade) Combined With Reinduction Chemotherapy in Children and Young Adults With Recurrent, Refractory or Secondary Acute Myeloid Leukemia
Brief Title: Bortezomib and Combination Chemotherapy in Treating Younger Patients With Recurrent, Refractory, or Secondary Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00323; U10CA098543 (NIH); CDR0000594224 (Registry Identifier: PDQ (Physician Data Query)); COG-AAML07P1 (Other: Children's Oncology Group); NCI-2009-00323 (Other: NCI)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myelomonocytic Leukemia (M4); Childhood Acute Basophilic Leukemia; Childhood Acute Eosinophilic Leukemia; Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Minimally Differentiated Myeloid Leukemia (M0); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Eosinophilic, Acute | interventions — Idarubicin; Cytarabine; Bortezomib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bortezomib 1.3mg/m2-assess efficacy-low anthracycline exposure (Experimental): Bortezomib 1.3mg/m2 to assess efficacy in low prior anthracycline exposure. Patients receive idarubicin IV (12 mg/m2/day) over 15 minutes on days 1-3, low-dose cytarabine IV (100 mg/m2/day) continuously over days 1-7, and bortezomib IV (1.3 mg/m2) on days 1, 4, and 8. All patients receive intrathecal cytarabine (30 mg - age 1-1.99 years, 50 mg - age 2-2.99 years, 70 mg - age ≥ 3 years) prior to courses 1 and 2. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity (closed as of 08/01/10). Dosage modification based on age < 3 years old.
  Interventions: Drug: idarubicin; Drug: cytarabine; Drug: bortezomib; Other: laboratory biomarker analysis
- Bortezomib 1.0mg/m2-assess feasibility high anthracycline exp (Experimental): Bortezomib 1.0 mg/m2 to assess feasibility in high prior anthracycline exposure. Patients receive etoposide IV (150 mg/m2/dose) over 1 hour on days 1-5, high-dose cytarabine IV (1000 mg/m2/dose) over 1 hour twice daily on days 1-5, and bortezomib IV (1.0 mg/m2) on days 1, 4, and 8. All patients receive intrathecal cytarabine (30 mg - age 1-1.99 years, 50 mg - age 2-2.99 years, 70 mg - age ≥ 3 years) prior to courses 1 and 2. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cytarabine; Drug: bortezomib; Drug: etoposide; Other: laboratory biomarker analysis
- Bortezomib 1.3 mg/m2-assess feasibility high anthracycline exp (Experimental): Bortezomib 1.3 mg/m2 to assess feasibility in high prior anthracycline exposure. Patients receive etoposide IV (150 mg/m2/dose) over 1 hour on days 1-5, high-dose cytarabine IV (1000 mg/m2/dose) over 1 hour twice daily on days 1-5, and bortezomib IV (1.3 mg/m2) on days 1, 4, and 8. All patients receive intrathecal cytarabine (30 mg - age 1-1.99 years, 50 mg - age 2-2.99 years, 70 mg - age ≥ 3 years) prior to courses 1 and 2. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity (dose-finding phase closed as of 10/10).
  Interventions: Drug: cytarabine; Drug: bortezomib; Drug: etoposide; Other: laboratory biomarker analysis
- Bortezomib 1.3 mg/m2-assess efficacy high anthracycline exp (Experimental): Bortezomib 1.3 mg/m2 to assess efficacy in high prior anthracycline exposure. Patients receive etoposide IV (150 mg/m2/dose) over 1 hour on days 1-5, high-dose cytarabine IV (1000 mg/m2/dose) over 1 hour twice daily on days 1-5, and bortezomib IV (1.3 mg/m2) on days 1, 4, and 8. All patients receive intrathecal cytarabine (30 mg - age 1-1.99 years, 50 mg - age 2-2.99 years, 70 mg - age ≥ 3 years) prior to courses 1 and 2. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: cytarabine; Drug: bortezomib; Drug: etoposide; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
  Arms: Bortezomib 1.3mg/m2-assess efficacy-low anthracycline exposure
Drug: cytarabine — Given IV or IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Bortezomib 1.0mg/m2-assess feasibility high anthracycline exp; Bortezomib 1.3 mg/m2-assess efficacy high anthracycline exp; Bortezomib 1.3 mg/m2-assess feasibility high anthracycline exp
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and best dose of bortezomib and to see how well it works when given together with combination chemotherapy in treating younger patients with recurrent, refractory, or secondary acute myeloid leukemia (AML). Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as idarubicin, cytarabine, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with bortezomib may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities and tolerability of bortezomib in combination with standard-relapse AML therapy (idarubicin/cytarabine or etoposide/high-dose cytarabine) in pediatric and young adult patients with relapsed or primary-refractory or secondary AML.

II. To estimate the complete response rate to the Arm A and Arm B regimens.

SECONDARY OBJECTIVES:

I. To determine whether bortezomib inhibits proteasome activity, NF-kB activity and induces apoptosis pathway proteins in leukemia myeloblasts. II. To determine the feasibility of measuring AML stem cells in relapsed and recovering bone marrow.

OUTLINE: This is a multicenter, dose-escalation study of bortezomib. Patients are stratified according to anthracycline*-equivalent cumulative exposure (≤ 400 mg/m² vs > 400 mg/m²). Patients are assigned to 1 of 2 groups.

GROUP I (efficacy phase, patients with ≤ 400 mg/m² anthracycline-equivalent cumulative exposure - Closed as of 08/01/10): Patients receive idarubicin IV over 15 minutes on days 1-3, low-dose cytarabine IV continuously over days 1-7, and bortezomib IV on days 1, 4, and 8.

GROUP II (dose-finding phase (closed as of 10/10) and efficacy phase, patients with > 400 mg/m² anthracycline*-equivalent cumulative exposure): Patients receive etoposide IV over 1 hour on days 1-5, high-dose cytarabine IV over 1 hour twice daily on days 1-5, and bortezomib IV on days 1, 4, and 8.

NOTE: * Anthracycline restriction no longer required for group 2 as of 10/02/10.

All patients receive intrathecal cytarabine prior to courses 1 and 2. In both arms, treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) according to WHO classification

  * At least 5% blasts in the bone marrow
  * With or without extramedullary disease
* To be eligible for the dose-finding phase (closed as of 10/10) :

  * Relapsed patients must meet the following criteria:

    * Must have had a prior diagnosis of AML, but may NOT have inv(16) or t(8;21) cytogenetics
    * May be in first or any subsequent relapse
    * If in first relapse, remission duration must be less than one year
  * Refractory patients must meet the following criteria:

    * Must have had a prior diagnosis of AML
    * May have received one or more attempt at remission induction
  * Patients with treatment-related AML may be previously treated or untreated for secondary AML
* To be eligible for the efficacy phase:

  * Relapsed patients must meet the following criteria:

    * Must have had a prior diagnosis of AML, with no restriction on prior cytogenetics
    * Must be in first relapse
    * Must not have received prior reinduction therapy
  * Refractory patients must meet the following criteria:

    * Must have had a prior diagnosis of AML
    * Must not have received more than one attempt at remission induction (which may consist of up to two therapy courses)
  * Patients with treatment-related AML must be previously untreated for secondary AML
* No juvenile myelomonocytic leukemia or acute promyelocytic leukemia (APL; FAB M3)
* Patients with the following CNS status are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia, such as cranial nerve palsy:

  * CNS 1, defined as absence of blasts in cerebral spinal fluid (CSF) on cytospin preparation, regardless of the number of WBCs
  * CNS 2, defined as presence of < 5/μL WBCs in CSF and cytospin positive for blasts, or > 5/uL WBCs but negative by Steinherz/Bleyer algorithm:

    * CNS 2a: < 10/μL RBCs; < 5/μL WBCs and cytospin positive for blasts
    * CNS 2b: ≥ 10/μL RBCs; < 5/μL WBCs and cytospin positive for blasts
    * CNS 2c: ≥ 10/μL RBCs; ≥ 5/μL WBCs and cytospin positive for blasts but negative by Steinherz/Bleyer algorithm
* Patients with CNS3 disease (presence of ≥ 5/μL WBCs in CSF and cytospin positive for blasts [in the absence of a traumatic lumbar puncture] and/or clinical signs of CNS leukemia) are not eligible
* CNS toxicity ≤ grade 2
* Lansky (patients ≤ 16 years of age) or Karnofsky (patients > 16 years of age) performance status (PS) 50-100%
* ECOG PS 0-2
* No Down syndrome
* No Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome
* No evidence of active graft-vs-host disease
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * 0.4 mg/dL for patients 1 month to < 6 months of age
  * 0.5 mg/dL for patients 6 months to < 1 year of age
  * 0.6 mg/dL for patients 1 to < 2 years of age
  * 0.8 mg/dL for patients 2 to < 6 years of age
  * 1 mg/dL for patients 6 to < 10 years of age
  * 1.2 mg/dL for patients 10 to < 13 years of age
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) for patients 13 to < 16 years of age
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) for patients ≥ 16 years of age
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* ALT < 3.0 times ULN for age (unless elevation due to leukemia involvement)
* Shortening fraction ≥ 27% by ECHO OR LVEF ≥ 50% by gated radionuclide
* Normal respiratory rate and pulse oximetry > 94% on room air
* FEV_1 ≥ 80% of predicted
* FVC and DLCO > 50% (corrected for hemoglobin)

  * Patients who are unable to perform pulmonary function tests (PFTs) (e.g., because of young age) will be excluded provided they have a medical history of significant prior pulmonary events or chronic pulmonary disease (e.g., pneumonia requiring mechanical ventilation support, pulmonary GVHD, pneumonectomy, or pulmonary toxin exposure)
  * Children with histories of resolved bronchiolitis, resolved viral pneumonias and well-controlled asthma are eligible, even if they are unable to perform PFTs
* Patients with seizure disorder may be enrolled if on a non-enzyme-inducing anticonvulsant and if seizures are well-controlled
* No uncontrolled infection
* No known allergy to idarubicin, cytarabine, etoposide, boron, mannitol or bortezomib
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Concurrent radiotherapy allowed for patients who present with a chloroma that is producing or threatens to produce an irreversible neurologic deficit
* Recovered from all prior chemotherapy, immunotherapy, or radiotherapy
* More than 2 weeks since prior cytotoxic chemotherapy (4 weeks for nitrosoureas), except for hydroxyurea, which is allowed up to 24 hours prior to first dose of study drug, and intrathecal chemotherapy, which is allowed immediately up to administration of study drug
* Prior steroid allowed as clinically indicated for patients with asthma

  * Hydrocortisone and methylprednisolone allowed as premedication in patients with a history of severe allergic reactions
* At least 7 days since prior biologic agents, such as steroids, retinoids, or donor lymphocyte infusion without conditioning
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 8 weeks since prior craniospinal radiotherapy or ≥ 50% radiation of pelvis
* At least 6 weeks since prior other bone marrow radiation
* At least 1 day since prior green tea containing products, any products containing vitamin C, flavanoids or other antioxidants (e.g., vitamins, herbal supplements), and foods with high vitamin C content
* No prior radiotherapy to > 25% of lung volume
* No prior total-body irradiation as part of a hematopoietic stem cell conditioning regimen
* At least 2 months since prior stem cell transplantation
* No concurrent graft-vs-host disease prophylactic medication
* No prior bortezomib or other proteasome inhibitors
* No other concurrent investigational drugs
* More than 4 days since prior growth factors that support platelet or white cell number or function
* No concurrent enzyme-inducing anticonvulsant medications known to be potent inducers of the cytochrome P450 system, including phenytoin, carbamazepine, and phenobarbital

  * Concurrent benzodiazepines and gabapentin allowed
* No concurrent grapefruit juice with bortezomib
* No other concurrent cancer chemotherapy or immunomodulating agents
* No concurrent corticosteroids as anti-emetic therapy

  * Concurrent corticosteroids therapy allowed as treatment or prophylaxis for anaphylactic reactions, symptoms of cytarabine syndrome, and as treatment for presumptive bortezomib-induced pulmonary toxicity.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Moscow, Principal Investigator — Children's Oncology Group
Locations (82):
- United States (77):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Miller Children's Hospital, Long Beach, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Childrens Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph Children's Hospital of Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Childrens Memorial Hospital, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University - Breslin Cancer Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical Center-Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UMDNJ - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Palmetto Health Richland, Columbia, South Carolina
  - Sanford University of South Dakota Medical Center, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (4):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Started | 18 | 6 | 6 | 22
Completed | 14 | 6 | 6 | 20
Not Completed | 4 | 0 | 0 | 2
Not completed — ineligible | 2 | 0 | 0 | 2
Not completed — inevaluable | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp | Total
Number analyzed (Participants) | 18 | 6 | 6 | 22 | 52
Age, Continuous [Mean (Standard Deviation); unit: days] | 4121.72 (2569.95) | 5637.0 (1757.39) | 2812.5 (1769.83) | 3365.0 (2227.99) | 3984.06 (2081.29)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 4 | 6 | 21 | 46
  Between 18 and 65 years | 3 | 2 | 0 | 1 | 6
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 4 | 13 | 30
  Male | 7 | 4 | 2 | 9 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 2 | 7
  White | 11 | 3 | 3 | 18 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 1 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 3 | 7
  Not Hispanic or Latino | 13 | 6 | 5 | 17 | 41
  Unknown or Not Reported | 2 | 0 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 17 | 5 | 6 | 20 | 48
  Canada | 1 | 1 | 0 | 1 | 3
  Australia | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Number of participants with dose limiting toxicity.
Time Frame: During Course 1
Measure: Number; unit: participants
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Number analyzed (Participants) | 14 | 6 | 6 | 20
participants | 0 | 1 | 0 | 0

2. Primary Outcome: Overall Response (Complete Remission [CR] and CR With Partial Recovery [CRp]) During Course 1
Description: Overall response (complete remission [CR] and CR with partial recovery [CRp]) during course 1.
Time Frame: After course 1
Measure: Number; unit: participants
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Number analyzed (Participants) | 14 | 6 | 6 | 20
participants | 4 | 2 | 2 | 9

3. Secondary Outcome: NF-kB Activity by Enzyme-linked Immunosorbent Assay (ELISA)
Description: NF-kB activity will be measured as a continuous variable (ng NF-kB/Mg protein). Differences in NF-κB activity between time points will be assessed using summary statistics such as mean, standard deviation, and range. We may perform exploratory analyses to determine if single time point measurements, or the difference between time points, correlate with treatment response.
Time Frame: At baseline, prior to and up to 24 hours after bortezomib treatment
Population: Ineligible patients (n=4) are excluded. Patients without available data (n=36) are excluded.
Measure: Mean (Standard Deviation); unit: ng/Mg protein
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Number analyzed (Participants) | 5 | 1 | 1 | 5
ng/Mg protein
  Baseline | 718.218 (418.149339) | 655.4 | 974.66 | 408.144 (484.084297)
  24 Hrs after treatment | 774.1925 (410.667711) | 345.46 | 855.96 | 497.31 (449.312899)

4. Secondary Outcome: Proteasome Inhibition Activity
Description: Mean and standard deviation of β1 and β5- Results are ratios (proteasome subunit/β-actin based on loading of 15 µg total protein, normalized to CEM).
Time Frame: At baseline
Population: Ineligible patients (n=4) are excluded. Patients without available data (n=36) are excluded. The data summarized are only at baseline as that is the only data available.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Number analyzed (Participants) | 4 | 1 | 0 | 7
ratio
  Baseline β1 | 0.08115 (0.0860893) | 0.7894 |  | 0.2895143 (0.2974052)
  Baseline β5 | 0.121575 (0.0691725) | 0.2576 |  | 0.3721286 (0.7140883)

5. Secondary Outcome: Protein Expression Assessed by Western Blot
Description: Relative expression of apoptotic and cell cycle proteins will be characterized using descriptive statistics. If differences are noted between pre and post-treatment protein expression, pairwise comparisons will be made using paired t-test or an equivalent nonparametric test if the data are non-normally distributed. The normality assumption will be assessed on the log-transformed data prior to paired t-test evaluation.
Time Frame: At baseline, prior to and up to 24 hours after bortezomib treatment
Population: These data will never be collected because the investigators decided not to perform quantitative biologic analysis.
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Feasibility of Stem Cell Quantitation: Percentage of Leukemia Initiation Cells (LIC) Depletion
Description: Descriptive statistics to assess mean +/- standard deviation for the percentage leukemia initiation cells (LIC) depletion.
Time Frame: At baseline and after completion of course 1
Population: Ineligible patients (n=4) are excluded. Patients without available data (n=42) are excluded.
Measure: Mean (Standard Deviation); unit: percentage of LIC depletion
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Number analyzed (Participants) | 3 | 0 | 1 | 2
percentage of LIC depletion
  Prior to Treatment | 0.013667 (0.02108) |  | 0.2 | 1.6385 (2.06887)
  Post Treatment | 0.021 (0.036373) |  | 0.43 | 0.0435 (0.0615183)

ADVERSE EVENTS:
Description: The ineligible patients are not included in the adverse event reporting.
Arm/Group | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp
Serious Adverse Events (participants affected / at risk) | 3/16 | 3/6 | 1/6 | 5/20
Other Adverse Events (participants affected / at risk) | 14/16 | 5/6 | 5/6 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure (N=16) | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp (N=6) | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp (N=6) | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Adeers submitted
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 1 — Adeers submitted
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 — Adeers submitted
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 — Adeers submitted
Anal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Adeers submitted
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 — Adeers submitted
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 — Adeers submitted
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1 — Adeers submitted
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Creatinine increased (Investigations) | 0 | 1 | 0 | 1 — Adeers submitted
Death NOS (General disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Adeers submitted
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 — Adeers submitted
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Adeers submitted
GGT increased (Investigations) | 0 | 1 | 0 | 1 — Adeers submitted
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 — Adeers submitted
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — Adeers submitted
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 — Adeers submitted
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 — Adeers submitted
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Adeers submitted
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 — Adeers submitted
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 — Adeers submitted
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 — Adeers submitted
Infections and infestations - Other, specify (Infections and infestations) | 0 | 2 | 0 | 1 — Adeers submitted
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 — Adeers submitted
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Adeers submitted
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 — Adeers submitted
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Adeers submitted
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — Adeers submitted
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 — Adeers submitted
Psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0 — Adeers submitted
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Adeers submitted
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 — Adeers submitted
Sepsis (Infections and infestations) | 0 | 1 | 0 | 2 — Adeers submitted
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bortezomib 1.3mg/m2-assess Efficacy-low Anthracycline Exposure (N=16) | Bortezomib 1.0mg/m2-assess Feasibility High Anthracycline Exp (N=6) | Bortezomib 1.3 mg/m2-assess Feasibility High Anthracycline Exp (N=6) | Bortezomib 1.3 mg/m2-assess Efficacy High Anthracycline Exp (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 — Adeers not subm
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 — Adeers not subm
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 — Adeers not subm
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 2 — Adeers not subm
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — Adeers not subm
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0 — Adeers not subm
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 0 — Adeers not subm
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 1 — Adeers not subm
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 — Adeers not subm
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 — Adeers not subm
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 — Adeers not subm
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 — Adeers not subm
Capillary leak syndrome (Vascular disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 2 — Adeers not subm
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Dysphasia (Nervous system disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 1 — Adeers not subm
Esophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Fatigue (General disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 2 | 2 | 5 — Adeers not subm
Fever (General disorders) | 0 | 0 | 0 | 4 — Adeers not subm
Fibrinogen decreased (Investigations) | 1 | 0 | 0 | 0 — Adeers not subm
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — Adeers not subm
GGT increased (Investigations) | 0 | 1 | 0 | 0 — Adeers not subm
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0 — Adeers not subm
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 — Adeers not subm
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3 | 2 | 3 — Adeers not subm
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 — Adeers not subm
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Infections and infestations - Other, specify (Infections and infestations) | 9 | 3 | 4 | 3 — Adeers not subm
INR increased (Investigations) | 1 | 0 | 0 | 0 — Adeers not subm
Investigations - Other, specify (Investigations) | 0 | 0 | 1 | 0 — Adeers not subm
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2 — Adeers not subm
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 — Adeers not subm
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 1 | 1 — Adeers not subm
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 2 — Adeers not subm
Neutrophil count decreased (Investigations) | 3 | 2 | 1 | 0 — Adeers not subm
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Pain (General disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 — Adeers not subm
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1 | 0 — Adeers not subm
Platelet count decreased (Investigations) | 1 | 1 | 1 | 0 — Adeers not subm
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 — Adeers not subm
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 — Adeers not subm
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 — Adeers not subm
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Adeers not subm
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — Adeers not subm
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 | 0 | 0 — Adeers not subm
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 1 — Adeers not subm
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2 — Adeers not subm
White blood cell decreased (Investigations) | 3 | 2 | 1 | 0 — Adeers not subm

LIMITATIONS AND CAVEATS:
The secondary outcome measure "Protein Expression Assessed by Western Blot" will never be reported as the investigators decided not to perform quantitative biologic analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less